CLINICAL TRIAL: NCT00216567
Title: A Randomized, Open Label, Comparative, Multi-center Clinical Trial to Determine the Efficacy and Safety of Topiramate Comparing With Carbamazepine in Benign Rolandic Epilepsy.
Brief Title: Safety and Efficacy of Topamax Versus Carbamazepine in Benign Rolandic Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005077
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Epilepsy, Rolandic
Keywords: Benign rolandic epilepsy; Topiramate
MeSH Terms: conditions — Epilepsy, Rolandic | interventions — Topiramate

INTERVENTIONS:
Drug: topamax

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Topiramate in comparison to Carbamazepine in Benign rolandic epilepsy.

DETAILED DESCRIPTION:
Benign rolandic epilepsy (BRE) is a common seizure disorder confined solely to children. The disorder is marked clinically by nocturnal generalized tonic-clonic seizures and diurnal seizures consisting of simple partial seizures consisting of brief unilateral facial clonic activity, dysphasia, and drooling. The EEG abnormalities are unique, consisting of generally high amplitude, centrotemporal spikes that are activated by sleep. The seizures typically begin in the first decade and almost always stop by age 16 years. The seizures are usually infrequent although clusters of seizures do occur. When the physician elects to treat, the seizures are usually easily controlled. This is a randomized, open label, active controlled, multi-center based clinical trial to determine the efficacy and safety of Topiramate comparing with Carbamazepine in Benign rolandic epilepsy. The study hypothesis is that topiramate will be more effective in treatment of Benign rolandic epilepsy than Carbamazepine, as evaluated by seizure-free rate at 24 weeks and Intellectual Functioning : KEDI-WISC (Korean Educational Development Institute Wechsler Intelligence Scale for Children-Revised) and is generally well-tolerated.

Topiramate (target dose) 4mg/kg/day, B.I.D, oral, for 24 weeks, carbamazepine(target dose) 30mg/kg/day, B.I.D, oral, for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose guardians submitted written consent
* Subjects with more than 2 seizures in last 1 year
* Subjects showing one of the following additional criteria
* Psychological burden due to seizure
* Seizure in daytime
* More than 3 seizures in last 6 month
* Convulsive seizure

Exclusion Criteria:

* Abnormalities on MRI, EEG
* Mental retardation
* History of seizure relapse
* Seizures due to organic causes
* Medically serious acute or chronic disease or progressive and degenerative disorders
* Patients who have received an investigational medication

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2002-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Seizure-free rate at 24 weeks in comparison of topiramate to carbamazepine

SECONDARY OUTCOMES:
In comparison of topiramate to carbamazepine, Intellectual Functioning : KEDI-WISC (Korean Educational Development Institute Wechsler Intelligence Scale for Children-Revised)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.